CLINICAL TRIAL: NCT04908111
Title: A Cancer Research UK Phase I/IIa Trial of Chimpanzee Adenovirus Oxford 1 (ChAdOx1) and Modified Vaccinia Ankara (MVA) Vaccines Against MAGE-A3 and NY-ESO-1 With Standard of Care Treatment (Chemotherapy and an Immune Checkpoint Inhibitor)
Brief Title: A Trial of ChAdOx1 and MVA Vaccines Against MAGE-A3 and NY-ESO-1
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor has decided to permanently close recruitment
Sponsor: Cancer Research UK (Other)
Collaborators: Vaccitech Oncology Ltd (VOLT) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/20/001; 2019-003015-64 (EudraCT Number)
Record Dates: First submitted 2021-04-23; First posted 2021-06-01 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); Squamous Oesophageal Cancer
Keywords: Immunotherapy; Vaccine; Cancer; Oncology; Lung Cancer; NSCLC Non-small cell lung cancer; Esophageal neoplasms; Neoplasms, Squamous Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Lung Neoplasms; Esophageal Neoplasms; Neoplasms, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Safety Run-In (Experimental): Six evaluable patients will receive the trial vaccines with Standard of Care (SoC) treatment to confirm they are safe before opening the next stage of the trial. These patients will not be randomised.
  Interventions: Biological: ChAdOx1-MAGEA3-NYESO (Route = IM injection, Dose = 5×10^10 vp); Biological: MVA-MAGEA3 (Route = IM injection, Dose = 1.3×10^8 pfu); Biological: MVA-NYESO (Route = IM injection, Dose = 1.5×10^8 pfu)
- NSCLC Arm A: Trial vaccines with SoC treatment (Experimental): Approximately 40 patients will be randomised to receive the trial vaccines with SoC treatment in this arm.
  Interventions: Biological: ChAdOx1-MAGEA3-NYESO (Route = IM injection, Dose = 5×10^10 vp); Biological: MVA-MAGEA3 (Route = IM injection, Dose = 1.3×10^8 pfu); Biological: MVA-NYESO (Route = IM injection, Dose = 1.5×10^8 pfu)
- NSCLC Arm B: SoC treatment (Other): Approximately 40 patients will be randomised to receive SoC treatment alone in this arm.
  Interventions: Combination Product: Standard of care treatment
- Squamous Oesophageal Cancer Cohort (Experimental): Approximately 17 patients with squamous oesophageal cancer will received the trial vaccines with SoC treatment
  Interventions: Biological: ChAdOx1-MAGEA3-NYESO (Route = IM injection, Dose = 5×10^10 vp); Biological: MVA-MAGEA3 (Route = IM injection, Dose = 1.3×10^8 pfu); Biological: MVA-NYESO (Route = IM injection, Dose = 1.5×10^8 pfu)

INTERVENTIONS:
Biological: ChAdOx1-MAGEA3-NYESO (Route = IM injection, Dose = 5×10^10 vp) — Patients commence their SoC chemotherapy in combination with an immune checkpoint inhibitor in 3 weekly cycles. Patients are screened during the first 2 cycles of SoC treatment to confirm eligibility for the trial.
  Patients who receive trial vaccines (safety run in stage, Arm A of the NSCLC randomisation cohort and Squamous Oesophageal Cancer Cohort) continue to receive their SoC treatment plus:
  * First prime ChAdOx1-MAGEA3-NYESO vaccine on Cycle 3 Day 1 of SoC treatment.
  * First boost MVA-MAGEA3 vaccine, and if applicable a first boost MVA-NYESO vaccine, 21 days later.
  * For patients who have not progressed: second prime ChAdOx1-MAGAEA3-NYESO vaccine 15 weeks following first prime vaccine
  * Second boost MVA-MAGAE3 vaccine, and if applicable a second boost MVA-NYESO vaccine, 21 days following second prime vaccine
  Patients in Arm B of the NSCLC randomisation cohort will continue to receive their SoC treatment only throughout the trial (i.e. no trial vaccines)
  Arms: NSCLC Arm A: Trial vaccines with SoC treatment; Safety Run-In; Squamous Oesophageal Cancer Cohort
Biological: MVA-MAGEA3 (Route = IM injection, Dose = 1.3×10^8 pfu) — Patients commence their SoC chemotherapy in combination with an immune checkpoint inhibitor in 3 weekly cycles. Patients are screened during the first 2 cycles of SoC treatment to confirm eligibility for the trial.
  Patients who receive trial vaccines (safety run in stage, Arm A of the NSCLC randomisation cohort and Squamous Oesophageal Cancer Cohort) continue to receive their SoC treatment plus:
  * First prime ChAdOx1-MAGEA3-NYESO vaccine on Cycle 3 Day 1 of SoC treatment.
  * First boost MVA-MAGEA3 vaccine, and if applicable a first boost MVA-NYESO vaccine, 21 days later.
  * For patients who have not progressed: second prime ChAdOx1-MAGAEA3-NYESO vaccine 15 weeks following first prime vaccine
  * Second boost MVA-MAGAE3 vaccine, and if applicable a second boost MVA-NYESO vaccine, 21 days following second prime vaccine
  Patients in Arm B of the NSCLC randomisation cohort will continue to receive their SoC treatment only throughout the trial (i.e. no trial vaccines)
  Arms: NSCLC Arm A: Trial vaccines with SoC treatment; Safety Run-In; Squamous Oesophageal Cancer Cohort
Combination Product: Standard of care treatment — Patients will continue to receive SoC treatment (chemotherapy and checkpoint inhibitor).
  Arms: NSCLC Arm B: SoC treatment
Biological: MVA-NYESO (Route = IM injection, Dose = 1.5×10^8 pfu) — Patients commence their SoC chemotherapy in combination with an immune checkpoint inhibitor in 3 weekly cycles. Patients are screened during the first 2 cycles of SoC treatment to confirm eligibility for the trial.
  Patients who receive trial vaccines (safety run in stage, Arm A of the NSCLC randomisation cohort and Squamous Oesophageal Cancer Cohort) continue to receive their SoC treatment plus:
  * First prime ChAdOx1-MAGEA3-NYESO vaccine on Cycle 3 Day 1 of SoC treatment.
  * First boost MVA-MAGEA3 vaccine, and if applicable a first boost MVA-NYESO vaccine, 21 days later.
  * For patients who have not progressed: second prime ChAdOx1-MAGAEA3-NYESO vaccine 15 weeks following first prime vaccine
  * Second boost MVA-MAGAE3 vaccine, and if applicable a second boost MVA-NYESO vaccine, 21 days following second prime vaccine
  Patients in Arm B of the NSCLC randomisation cohort will continue to receive their SoC treatment only throughout the trial (i.e. no trial vaccines)
  Arms: NSCLC Arm A: Trial vaccines with SoC treatment; Safety Run-In; Squamous Oesophageal Cancer Cohort

SUMMARY:
This clinical trial is looking at two new vaccines called ChAdOx1-MAGEA3-NYESO, MVA-MAGEA3 and MVA-NYESO given with patients' standard of care treatment (chemotherapy and an immune checkpoint inhibitor).

DETAILED DESCRIPTION:
Patients with non-small cell lung cancer (NSCLC) or squamous oesophageal cancer will be entered into the trial as these tumour types are commonly known to have MAGE-A3 and NY-ESO-1 proteins on their cancer cells. The vaccines contain harmless parts of these proteins allowing them to show these proteins to the immune system. It is expected the immune system will 'learn' that these proteins are foreign to the body. The immune system should then attack the proteins on the cancer cells, killing them. It is expected the vaccines will help the chemotherapy and immune checkpoint inhibitor to work better.

This is a first-in-human clinical trial which has two stages:

* A 'Safety Run In' stage where six evaluable patients will receive the trial vaccines with standard of care treatment to confirm they are safe before opening the next stage.
* A 'Rolling Recruitment' stage consisting of two cohorts:

  1. NSCLC Randomisation Cohort of approximately 80 patients with NSCLC will be randomly allocated by computer (randomised) to one of two groups (arms). Patients in Arm A will receive the vaccines with their standard of care treatment and patients in Arm B will continue with their standard of care treatment alone. There is a 1 in 2 chance patients will receive the vaccines.
  2. Squamous Oesophageal Cancer Cohort: Approximately 17 patients with squamous oesophageal cancer will be recruited to receive trial vaccines with their standard of care treatment.

The main aims of the trial are to find out:

* More about potential side effect of the vaccine and how they can be managed.
* Whether the vaccines with standard of care treatment are better at shrinking NSCLC than just the standard of care treatment alone.
* What happens to the vaccines inside the body.

ELIGIBILITY:
Inclusion Criteria

1. Written (signed and dated) informed consent for both pre-screening and the main trial and capable of co-operating with any investigational medicinal product (IMP) administration and follow-up.
2. Histologically or cytologically proven Stage IIIB, IIIC or IV squamous NSCLC or Stage IIIB or IV non-squamous NSCLC scheduled to receive pembrolizumab and chemotherapy as SoC at the time of enrolment or randomisation. Patients can receive up to two cycles of SoC pembrolizumab in combination with chemotherapy prior to enrolment or randomisation to the trial.

   Or histologically proven inoperable Stage III or IV squamous cell carcinomas of the oesophagus or gastro-oesophageal junction (referred to as squamous oesophageal cancer) scheduled to receive or continue to receive chemotherapy and pembrolizumab as SoC at the time of enrolment.
3. NSCLC patients with no prior immune checkpoint inhibitor therapy prior to the pembrolizumab they are receiving in combination with chemotherapy at time of enrolment or randomisation.

   1. For non-squamous NSCLC patients, the patient has not received previous systemic therapy for advanced/metastatic disease. Completion of treatment for earlier stage disease with chemotherapy with or without radiotherapy as part of neoadjuvant/radical/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of recurrent locally advanced or metastatic disease.
   2. For squamous NSCLC patients, the patient has not received previous cytotoxic chemotherapy for advanced/metastatic disease. Completion of treatment for earlier stage disease with chemotherapy with or without radiotherapy as part of neoadjuvant/radical/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of recurrent locally advanced or metastatic disease.

   Or patients with squamous oesophageal cancer with no prior systemic therapy for advanced disease and with no prior immune checkpoint inhibitor therapy prior to the chemotherapy and immune checkpoint inhibitor they are receiving at time of enrolment to the trial. Completion of treatment for earlier stage disease with chemotherapy with or without radiotherapy as part of neoadjuvant/radical/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of recurrent locally advanced or metastatic disease.
4. Have at least one measurable lesion according to RECIST v1.1. Note: A measurable lesion may be biopsied at screening and on trial, however that lesion cannot be selected as a target lesion for disease assessment according to RECIST v1.1.
5. Confirmed PD-L1 status (tumour proportion score) for NSCLC patients. Or a confirmed PD-L1 combined positive score for patients with squamous oesophageal cancer.
6. Archival tumour tissue or new biopsy expressing MAGE-A3 as demonstrated by quantitative Reverse Transcription Polymerase Chain Reaction (RT-qPCR).
7. Life expectancy of at least 12 weeks.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. Haematological and biochemical indices within the ranges shown below. These measurements should be performed to confirm the patient's eligibility.

   Haemoglobin ≥90 g/L

   Absolute neutrophil count ≥1.5×10^9/L (growth factor support Granulocyte-Colony Stimulating Factor is allowed when used as part of routine supportive therapy for SoC)

   Platelet count ≥100×10^9/L

   International normalized ratio (INR) ≤1.5* AND prothrombin time (PT) OR Activated partial thromboplastin time (aPTT) ≤1.5* × Upper Limit of Normal (ULN) *unless participant is receiving anticoagulant therapy as long as INR or PT/aPTT is within therapeutic range of intended use of anticoagulants.

   Bilirubin ≤1.5 × ULN OR <3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia)

   Alanine aminotransferase or aspartate aminotransferase ≤3.0 × ULN OR ≤5.0 × ULN in presence of liver metastases

   Calculated creatinine clearance (using the Cockcroft & Gault [C&G] formula) ≥50 mL/min or serum creatinine ≤1.5 × ULN
10. Aged 18 years or over at the time pre-screening consent is given.

Exclusion Criteria

1. For non-squamous NSCLC patients, patients who have received previous systemic therapy for advanced/metastatic disease prior to the pembrolizumab they are receiving in combination with chemotherapy at time of enrolment or randomisation. Completion of treatment for earlier stage disease with chemotherapy with or without radiotherapy as part of neoadjuvant/radical/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of recurrent locally advanced or metastatic disease. Palliative radiotherapy is allowed. Irradiated lesions will not be evaluable for response.

   For squamous NSCLC patients, patients who have received previous cytotoxic chemotherapy for advanced/metastatic disease prior to the pembrolizumab they are receiving in combination with chemotherapy at time of enrolment or randomisation. Completion of treatment for earlier stage disease with chemotherapy with or without radiotherapy as part of neoadjuvant/radical/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of recurrent locally advanced or metastatic disease. Palliative radiotherapy is allowed. Irradiated lesions will not be evaluable for response.

   Or for patients with squamous oesophageal cancer - patients who have previously received systemic therapy for advanced disease and with no prior immune checkpoint inhibitor therapy prior to the SoC treatment outlined in this clinical trial. Completion of treatment for earlier stage disease with chemotherapy with or without radiotherapy as part of neoadjuvant/radical/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of recurrent locally advanced or metastatic disease. Palliative radiotherapy is allowed. Irradiated lesions will not be evaluable for response.
2. Previous therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T cell receptor (e.g., anti-CTLA-4, OX 40, anti-CD137). This does not include the immune checkpoint inhibitor patients receive in combination with chemotherapy commencing during screening prior to enrolment or randomisation to the trial.
3. Current or prior malignancy which could affect safety or efficacy assessment of the IMP or compliance with the protocol or interpretation of results. Patients with curatively-treated non-melanoma skin cancer, non-muscle-invasive bladder cancer, or carcinomas-in-situ are eligible.
4. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with symptomatically active brain metastases or leptomeningeal metastases. Patients with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during trial screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
5. Women of child-bearing potential (or are already pregnant or lactating). However, those patients who meet the following points are considered eligible:

   * Have a negative serum or urine pregnancy test before enrolment or randomisation and;
   * Agree to use two forms of contraception (one effective form plus a barrier method) [oral, injected or implanted hormonal contraception and condom; intra-uterine device and condom; diaphragm with spermicidal gel and condom] or agree to sexual abstinence, effective from the first administration of ChAdOx1-MAGEA3-NYESO, throughout the treatment phase of the trial and for 6 months afterwards.
6. Male patients with partners of child-bearing potential. However, those patients who meet the following points are considered eligible:

   * They agree to take measures not to father children by using a barrier method of contraception (condom plus spermicide) or to sexual abstinence effective from the Cycle 3 Day 1 of SoC treatment, throughout the treatment phase of the trial and for six months afterwards.
   * Men with partners of child-bearing potential must also be willing to ensure that their partner uses an effective method of contraception for the same duration for example, hormonal contraception, intra-uterine device, diaphragm with spermicidal gel or sexual abstinence.
   * Men with pregnant or lactating partners must be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure to the foetus or neonate.
7. Major thoracic or abdominal surgery from which the patient has not yet recovered. Patients who have undergone other types of surgery which the Chief Investigator and Sponsor agree would not compromise patient safety on trial are eligible.
8. Electrocardiogram (ECG) with clinically significant abnormalities or with QTcF interval (QT corrected using Fridericia's formula) >480 msec.
9. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
10. Historically known to be serologically positive for hepatitis B or human immunodeficiency virus (HIV). Patients with previous Hepatitis C exposure but no current infection are eligible to participate.
11. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
12. Has received COVID-19 Vaccine AstraZeneca (previously named AZD1222 or ChAdOx1-nCoV-19) vaccine within six weeks of commencing chemotherapy and an immune checkpoint inhibitor.
13. Has received any other live vaccination within four weeks before enrolment or randomisation to the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
14. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug. Use of short (<7 day) courses of steroids as part of the SoC treatment management is allowed.
15. Has undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years. Participants who have had a transplant greater than 5 years ago are eligible as long as there are no symptoms of graft versus host disease.
16. Has previously experienced severe hypersensitivity (greater than or equal to Grade 3) to an immune checkpoint inhibitor, ChAdOx1 or MVA vaccines and/or any of their excipients.
17. History of a severe allergy to eggs or history of severe allergic reaction to any previous vaccination.
18. History of heparin-induced thrombocytopenia and thrombosis.
19. History of Capillary Leak Syndrome.
20. Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase I/IIa trial. Participation in an observational trial or interventional clinical trial which does not involve administration of an IMP and which would not place an unacceptable burden on the patient in the opinion of the Investigator and Medical Advisor would be acceptable.
21. Any other condition, which in the Investigator's opinion, would not make the patient a good candidate for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2029-03-06 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of the trial vaccines with SoC treatment (chemotherapy and an immune checkpoint inhibitor). | From time of written consent to participate in the trial until the End of Treatment visit for each patient. Any trial vaccine-related serious adverse events that become known after this period will be reported up to the end of trial (Max 89 Months).
  Incidence of adverse events (including injection site reactions and toxicity), including relatedness, seriousness and severity (graded according to the National Cancer Institute - Common Terminology Criteria for Adverse Events [NCI-CTCAE] Version 5.0).

SECONDARY OUTCOMES:
To determine the efficacy (Progression Free Survival [PFS], in months) of the trial vaccines when given with SoC treatment (chemotherapy and immune checkpoint inhibitor). | Until end of efficacy and survival follow-up (Max 5 years) for non-vaccinated patients and end of extended follow-up (Max 89 months) for vaccinated patients.
  PFS will be assessed as time from Cycle 3 Day 1 of SoC treatment to the date of disease progression. using Response Evaluation Criteria in Solid Tumours (RECIST) and immune RECIST (iRECIST).
To determine the efficacy (Overall Response Rate [ORR], in months) of the trial vaccines when given with SoC treatment (chemotherapy and immune checkpoint inhibitor). | Until end of efficacy and survival follow-up (max 5 years) for non-vaccinated patients and end of extended follow-up (Max 89 months) for vaccinated patients.
  ORR will be reported as the number of randomised patients who have achieved a complete response or partial response.
To determine the efficacy (Overall Survival [OS], in months) of the trial vaccines when given with SoC treatment (chemotherapy and immune checkpoint inhibitor). | Until end of efficacy and survival follow-up (Max 5 years) for non-vaccinated patients and end of extended follow-up (Max 89 months) for vaccinated patients.
  OS will be assessed as time from Cycle 3 Day 1 of SoC treatment to the date of death from any cause.
To determine the immunogenicity (antigen-specific peripheral response) of the trial vaccines given with SoC treatment (chemotherapy and an immune checkpoint inhibitor). | Screening (prior to commencing SoC treatment, Cycle 3 Day 1 (each cycle is 21 days), Cycle 3 Day 15/2 weeks after ChAdOx1-MAGEA3-NYESO vaccination, Cycle 4 Day 1, Cycle 4 Day 7/1 week after MVA vaccination and at End of Treatment visit (Max 40 weeks).
  Percentage of patients showing peripheral immune response. Immunological response will be measured in patient blood by antigen-specific T cells by ex vivo ELISpot assay.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Blackhall, Prof, Principal Investigator — The Christie NHS Foundation Trust
Locations (9):
- United Kingdom (9):
  - Blackpool Victoria Hospital, Blackpool
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Guy's and St Thomas' NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Churchill Hospital, Oxford
  - Royal Preston Hospital, Preston
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified participant data that underlie the results reported on a publicly accessible database (text, figures, tables and supplementary information) will be shared with Cancer Research UK funded/ employed researchers whose proposed use of the data is approved by a review committee of the sponsor. All requests made within 5 years from the end of trial will be considered; requests made subsequently will be considered where possible. Data sharing requests should be sent to: drugdev@cancer.org.uk.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All requests made within 5 years from the end of trial will be considered; requests made subsequently will be considered where possible.
Access Criteria: Researchers who are funded or employed by Cancer Research UK whose proposed use of the data is approved by a review committee of CDD.
URL: https://www.cancerresearchuk.org/about-cancer/find-a-clinical-trial/a-trial-looking-at-a-vaccine-chemotherapy-and-an-immunotherapy-for-non-small-cell-lung-cancer-and-squamous-oesophageal-cancer?advagg=0